CLINICAL TRIAL: NCT01834729
Title: Effect of Stress and a Alpha-1 Antagonist on Anorectal Functions
Brief Title: Effects of Alpha-1 Antagonist, Stress and Relaxation on Anorectal Functions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Adil Bharucha, PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12-006090; 1UL1RR024150 (NIH); R01DK078924 (NIH)
Record Dates: First submitted 2013-04-15; First posted 2013-04-18 (Estimated); Results first posted 2019-01-11 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alfuzosin (Experimental): In Part A, subjects randomized to this arm will receive a single dose of oral alfuzosin immediate release (IR) 2.5 mg.
  In Part B, only constipated patients will receive oral alfuzosin (10 mg extended release (ER)) capsules.
  Interventions: Drug: Alfuzosin
- Placebo (Placebo Comparator): Subjects randomized to this arm will receive a single placebo capsule identical to the study drug.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Alfuzosin — oral alfuzosin immediate release (IR) 2.5 mg (Part A) or oral alfuzosin extended release (ER) 10 mg (Part B)
  Other Names: Xatral (immediate release 2.5 mg); Uroxatral (extended release 10 mg)
  Arms: Alfuzosin
Other: Placebo — placebo capsule identical to the study drug
  Arms: Placebo

SUMMARY:
This study is designed to better understand the effects of effects of stress, relaxation, and a medication alfuzosin on bowel control and emptying in healthy people and patients with bowel problems.

DETAILED DESCRIPTION:
Normally, bowel emptying requires relaxation of the anal sphincter (i.e., lowermost end of intestinal tract) and pelvic muscles. Some people cannot relax these muscles normally and experience constipation. Alfuzosin is a medication which is approved to treat bladder but not bowel problems.

ELIGIBILITY:
Inclusion criteria for controls (Part A only):

* Healthy
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Inclusion criteria for patients (Parts A and B):

* Women with chronic constipation for 1 year with any 2 or more of the following symptoms for 3 months or longer, i.e. <3 bowel motions/week, straining ≥ 25% of time, hard or lumpy stools ≥ 25% of time, incomplete evacuation ≥ 25% of time, feeling of anorectal blockage ≥ 25% of time.
* Able to provide written informed consent before participating in the study
* Able to communicate adequately with the investigator and to comply with the requirements for the entire study.

Exclusion criteria for controls (Part A); Items indicated with an asterisk (*) are also exclusion criteria for patients (Parts A and B):

* Clinical evidence of significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other disease that may interfere with the objectives of the study and/or pose safety concerns.*
* Current symptomatic orthostatic hypotension or history of hypotensive response as defined by a reduction of ≥ 30 mmHg in systolic or ≥ 20 mmHg in diastolic blood pressure.*
* Current symptoms of a functional gastrointestinal disorder assessed by questionnaire.
* Putative risk factors for pelvic floor trauma, i.e. six or more vaginal deliveries, birthweight >4500gms (macrosomia), or known 4th degree perineal tear.
* Inability to withdraw medications prior to the baseline period and throughout the study (except as protocol defined rescue medications):

  1. Medications that substantially alter GI transit* including laxatives, magnesium and aluminum containing antacids, prokinetics, erythromycin, narcotics, anti-cholinergics, tricyclic antidepressants, serotonin-norepinephrine reuptake inhibitors (SNRI) and newer antidepressants
  2. Selective serotonin reuptake inhibitor (SSRI) antidepressants are permissible at low, stable doses. All medications shall be reviewed and dis/approved by the principal investigator on a case by case basis.*
  3. Potent Cytochrome P450 3A4 (Cyp3A4) inhibitors such as ketoconazole, itraconazole and ritonavir, nitrates and phosphodiesterase inhibitors.* Note: stable doses of thyroid replacement, estrogen replacement, low dose aspirin for cardioprotection, and birth control (but with adequate backup contraception as drug-interactions with birth control have not been conducted) are permissible.*
* Stable dose of thyroxine will be permitted*
* Prolonged Q-Tc interval > 500 msec on ECG within the last three months*
* Estimated glomerular filtration rate (eGFR) < 60 mL/minute. * Based on guidelines and recommendations from the National Kidney Disease Education Program (NKDEP) of the National Institutes of Health (NIH) and the Kidney Disease Outcomes Quality Initiative (KDOQI) of the National Kidney Foundation, the an eGFR using the Modification of Diet in Renal Disease (MDRD) Study equation is more accurate than a creatinine clearance calculated from serum and urine measurements. The formula is eGFR (mL/min/1.73 m2) = 175 x (Scr)-1.154 x (Age)-0.203 x (0.742 if female) x (1.210 if African American). Based on our extensive experience in clinical practice and research studies, it is anticipated that all potentially eligible participants will have normal serum creatinine.
* History of allergies to alpha-1 adrenoreceptor antagonist*
* Active rectal inflammation, cancer; perianal sepsis; history of pelvic radiation, rectosigmoid surgery or inflammatory bowel disease*
* Pregnant women, prisoners and institutionalized individuals*
* Persons with a latex allergy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Result] Chakraborty S, Feuerhak K, Muthyala A, Harmsen WS, Bailey KR, Bharucha AE. Effects of Alfuzosin, an alpha1-Adrenergic Antagonist, on Anal Pressures and Bowel Habits in Women With and Without Defecatory Disorders. Clin Gastroenterol Hepatol. 2019 May;17(6):1138-1147.e3. doi: 10.1016/j.cgh.2018.08.036. Epub 2018 Aug 18. PMID 30130627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 38 healthy subjects and 36 subjects with constipation for 1 year or longer participated in the study. Both the healthy subjects and constipation subjects participated in Part A. Only the constipation subjects participated in Part B.
Groups:
- Control Placebo: Healthy subjects defined as not having a functional bowel disorder randomized to this arm will receive a placebo capsule identical to the study drug. Placebo: placebo capsule identical to the study drug.
- Control Alfuzosin: Healthy subjects defined as not having a functional bowel disorder randomized to this arm will receive a receive a single dose of oral alfuzosin immediate release (IR) 2.5 mg.
- Constipation Placebo: Subjects with constipation for 1 year or longer randomized to this arm will receive a placebo capsule identical to the study drug. Placebo: placebo capsule identical to the study drug
- Constipation Alfuzosin: Subjects with constipation for 1 year or longer randomized to this arm will receive a single dose of oral alfuzosin immediate release (IR) 2.5 mg.
Period: Overall Study
Arm/Group | Control Placebo | Control Alfuzosin | Constipation Placebo | Constipation Alfuzosin
Started | 18 | 20 | 18 | 18
Completed | 17 | 19 | 15 | 16
Not Completed | 1 | 1 | 3 | 2
Not completed — Did not return bowel diaries | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Control Placebo; Constipation Placebo: Subjects randomized to this arm will receive a placebo capsule identical to the study drug.
  Placebo: placebo capsule identical to the study drug
- Control Alfuzosin: Subjects randomized to this arm will receive a single dose of oral alfuzosin immediate release (IR) 2.5 mg.
- Constipation Alfuzosin: In this arm, only constipated patients will receive oral alfuzosin (10 mg extended release (ER)) capsules.
  Alfuzosin: oral alfuzosin immediate release (IR) 2.5 mg (Part A) or oral alfuzosin extended release (ER) 10 mg (Part B)
- Total: Total of all reporting groups
Arm/Group | Control Placebo | Control Alfuzosin | Constipation Placebo | Constipation Alfuzosin | Total
Number analyzed (Participants) | 18 | 20 | 18 | 18 | 74
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: A total of 38 healthy subjects and 36 subjects with constipation for 1 year or longer participated in the study. Both the healthy subjects and constipation subjects participated in Part A. Only the constipation subjects participated in Part B.
  years | 32 [26 to 51] | 45 [28 to 53] | 36 [26 to 50] | 40 [35 to 44] | 40 [26 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 20 | 18 | 18 | 74
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 18 | 18 | 74
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] — Population: A total of 38 healthy subjects and 36 subjects with constipation for 1 year or longer participated in the study. Both the healthy subjects and constipation subjects participated in Part A. Only the constipation subjects participated in Part B.
  kg/m^2 | 24 [24 to 29] | 27 [23 to 29] | 25 [21 to 30] | 25 [19 to 29] | 26 [23 to 29]

OUTCOME MEASURES:

1. Primary Outcome: Weekly Rate of Spontaneous Bowel Movements at 4 Weeks
Description: A bowel movement is considered a spontaneous bowel movement (SBM) if no laxative, enema, or suppository was taken in the preceding 24 hours.
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: spontaneous bowel movements per week
Groups:
- Constipation Alfuzosin: Constipated patients will receive oral alfuzosin (10 mg extended release (ER) capsules.
Arm/Group | Control Placebo | Control Alfuzosin | Constipation Placebo | Constipation Alfuzosin
Number analyzed (Participants) | 18 | 20 | 18 | 18
spontaneous bowel movements per week | 1.6 (0.3) | 1.3 (0.1) | 1.6 (0.4) | 1.3 (0.1)
Statistical Analysis 1: Comparison: Constipation Placebo vs Constipation Alfuzosin; Test type: Superiority; p = 0.78, Least squares means

2. Primary Outcome: Weekly Rate of Complete Spontaneous Bowel Movements at 4 Weeks
Description: If the subject indicates that the spontaneous bowel movement (SBM) was associated with a sensation of complete bowel emptying, the SBM will be counted as a complete spontaneous bowel movement (CSBM).
Time Frame: 4 weeks
Measure: Mean (Standard Error); unit: complete SBM per week
Groups:
- Constipation Alfuzosin: Constipated patients will receive oral alfuzosin (10 mg extended release (ER)) capsules.
Arm/Group | Control Placebo | Control Alfuzosin | Constipation Placebo | Constipation Alfuzosin
Number analyzed (Participants) | 18 | 20 | 18 | 18
complete SBM per week | 0.6 (0.1) | 0.7 (0.05) | 0.7 (0.1) | 0.7 (0.1)
Statistical Analysis 1: Comparison: Constipation Placebo vs Constipation Alfuzosin; Test type: Superiority; p = 0.57, Least squares means

ADVERSE EVENTS:
Time Frame: Subject safety monitoring was performed for six hours after treatment in healthy patients and two weeks in constipated patients.
Groups:
- Constipation Afluzosin: Constipated patients will receive oral alfuzosin (10 mg extended release (ER)) capsules.
Arm/Group | Control Placebo | Control Alfuzosin | Constipation Placebo | Constipation Afluzosin
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 1/20 | 1/18 | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Placebo (N=18) | Control Alfuzosin (N=20) | Constipation Placebo (N=18) | Constipation Afluzosin (N=18)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal cramps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Men were not studied; baseline bowel diary was not preceded by a run-in period; treatment phase only lasted 2 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-20): https://cdn.clinicaltrials.gov/large-docs/29/NCT01834729/Prot_SAP_000.pdf